CLINICAL TRIAL: NCT05162833
Title: Evaluation of the TheraNova Neuromodulation System to Provide Durable Relief of Overactive Bladder Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Theranova, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRD-10-1332
Record Dates: First submitted 2021-11-23; First posted 2021-12-17 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Maintenance group (Experimental): Subjects that completed the clinical study "Evaluation of the TheraNova Neuromodulation System for the Treatment of Overactive Bladder Symptoms" that were in the active treatment group will be offered to extend treatment for 3 months.
  Interventions: Device: TheraNova Neuromodulation Device

INTERVENTIONS:
Device: TheraNova Neuromodulation Device — TENS device

SUMMARY:
To evaluate the safety and durability of the TheraNova Neuromodulation System in overactive bladder (OAB) patients.

ELIGIBILITY:
Inclusion Criteria:

* Individual completed the clinical study "Evaluation of the TheraNova Neuromodulation System for the Treatment of Overactive Bladder Symptoms" (Protocol Number CRD-10-1330-01) as a subject in the Active Treatment group

  * Individual has at least ≥4 incontinence events with associated moderate or severe urgency (UUI events), with at least one UUI event per day, as recorded in the baseline 3-day voiding diary at week 0 of the clinical study "Evaluation of the TheraNova Neuromodulation System for the Treatment of Overactive Bladder Symptoms" (Protocol Number CRD-10- 1330-01)
  * Individual is ambulatory and able to use the toilet independently
  * Individual has not taken antimuscarinics, anticholinergics, beta-3 agonists, alpha blockers, 5-alpha reductase inhibitors, vasopressin analogues, tricyclic antidepressants, or phenazopyridine for at least 2 weeks prior to enrollment
  * Individual is not taking diuretics or has been on a steady dose of diuretics for at least 3 months
  * Individual is able to provide informed consent
  * Individual is capable and willing to follow all study-related procedures

Exclusion Criteria:

* Individual has recurrent UTI defined as ≥4 UTIs in the past 12 months

  * Female of childbearing age (≤50 years old) who is pregnant as confirmed by urine pregnancy test, or who plans to become pregnant during the study period
  * Individual has peripheral arterial disease
  * Individual has the presence of a urinary fistula, bladder stone, or interstitial cystitis
  * Individual has a diagnosis of prostate, urethral, or bladder cancer
  * Individual has morbid obesity (BMI ≥ 40)
  * Individual has clinically significant urethral stricture disease or bladder neck contracture
  * Individual has a metallic implant that is exposed above the bone surface (e.g. a bone fracture fixation plate, but not an embedded bone screw) and is located under the skin on the bottom of the foot for either foot or under the skin on the anterior aspect of the mid-thigh for either leg.
  * Individual has an implanted electrical and/or neurostimulator device (e.g. pacemaker, defibrillator, vagal neurostimulator, deep brain stimulator, spinal stimulator, sacral stimulator, bone growth stimulator, or cochlear implant)
  * Individual has been treated with percutaneous tibial nerve stimulation or pelvic floor muscle stimulation
  * Individual has been treated with onabotulinumtoxinA in the past 9 months
  * Individual has a clinically significant peripheral neuropathy
  * Individual has a history of pelvic pain as primary diagnosis in the past 12 months (VAS score of >4 (scale of 0 to 10)) Individual has neurogenic bladder (i.e. Multiple Sclerosis, Parkinson's, Spinal Cord Injury)
  * Individual has used an investigational drug, biologic, or medical device in the past 4 weeks
  * Individual is deemed unsuitable for enrollment in the study by the investigator based on the subject's history or physical examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-02-20 (Actual); Primary Completion 2023-12-08 (Actual); Study Completion 2023-12-08 (Actual)

PRIMARY OUTCOMES:
UUIs | 12 weeks
  change in the mean number of urge urinary incontinence (UUI) episodes per day from week 12 to week 24 (this study starts at 12 weeks)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - UC Davis Health, Sacramento, California
  - Stanford University Medical Center, Stanford, California

IPD SHARING:
Plan to Share IPD: Undecided